CLINICAL TRIAL: NCT02573233
Title: An Exploratory, Double-blind, Placebo-controlled Study of the Effects of Dupilumab on Airway Inflammation of Adults With Persistent Asthma
Brief Title: Evaluation of Dupilumab's Effects on Airway Inflammation in Patients With Asthma
Acronym: EXPEDITION
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PDY14192; 2015-001572-22 (EudraCT Number); U1111-1170-7168 (Other: UTN)
Record Dates: First submitted 2015-10-08; First posted 2015-10-09 (Estimated); Results first posted 2019-01-28 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — dupilumab; Fluticasone-Salmeterol Drug Combination; Budesonide; Formoterol Fumarate; Budesonide, Formoterol Fumarate Drug Combination; Mometasone Furoate; Mometasone Furoate, Formoterol Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo (for dupilumab), 2 subcutaneous injections on Day 1 (Week 1) as a loading dose followed by a single injection q2w from Week 2 to Week 14, added to stable inhaled corticosteroid/ long-acting beta-agonist (ICS/LABA) therapy. Salbutamol/albuterol or Levosalbutamol/levalbuterol was given as reliever medication.
  Interventions: Drug: Placebo; Drug: fluticasone propionate and salmeterol; Drug: budesonide and formoterol; Drug: mometasone furoate and formoterol
- Dupilumab (Experimental): Dupilumab, 2 subcutaneous injections on Day 1 as a loading dose for a total of 600 mg, followed by a single 300 mg injection q2w from Week 2 to Week 14, added to stable ICS/LABA therapy. Salbutamol/albuterol or Levosalbutamol/levalbuterol was given as reliever medication.
  Interventions: Drug: Dupilumab SAR231893/REGN668; Drug: fluticasone propionate and salmeterol; Drug: budesonide and formoterol; Drug: mometasone furoate and formoterol

INTERVENTIONS:
Drug: Placebo — Pharmaceutical form:solution Route of administration: subcutaneous
  Arms: Placebo
Drug: Dupilumab SAR231893/REGN668 — Pharmaceutical form:solution Route of administration: subcutaneous
  Arms: Dupilumab
Drug: fluticasone propionate and salmeterol — Pharmaceutical form:inhalation aerosol, inhalation powder Route of administration: inhaled
  Other Names: Advair
Drug: budesonide and formoterol — Pharmaceutical form:inhalation aerosol Route of administration: inhaled
  Other Names: Symbicort
Drug: mometasone furoate and formoterol — Pharmaceutical form:inhalation aerosol Route of administration: inhaled
  Other Names: Dulera

SUMMARY:
Primary Objective:

To evaluate the effect of dupilumab, compared to placebo, on airway inflammation in participants with persistent asthma.

Secondary Objective:

To assess the safety, tolerability, and immunogenicity of dupilumab compared to placebo.

DETAILED DESCRIPTION:
The total study duration for each participant was between approximately 29 and maximum of 30 weeks, consisting of a screening period of 5 weeks and optional up to 7 additional days, a treatment period of 12 weeks, and a post-treatment period of 12 weeks.

Participants who completed the treatment period could be eligible to participate in an open-label extension study.

ELIGIBILITY:
Inclusion criteria:

* Male and female adults with a physician diagnosis of persistent asthma for ≥12 months.
* Existing treatment with medium to high dose inhaled corticosteroids in combination with a long-acting beta agonist for at least 3 months with a stable dose ≥1 month prior to Visit 1 (Screening Visit).
* Treatment with a third asthma controller for at least 3 months with a stable dose >=1 month prior to Visit 1 was allowed.
* Pre-bronchodilator forced expiratory volume (FEV1) 55 to 85% of predicted normal.

Exclusion criteria:

* Participants <18 years or >65 years.
* Fractional exhaled nitric oxide (FeNO) <26 parts per billion (ppb) at Visit 1 (Screening Visit).
* Chronic obstructive pulmonary disease or other lung diseases (eg, idiopathic pulmonary fibrosis, eosinophilic granulomatosis with polyangiitis [Churg-Strauss Syndrome]) which could impair lung function.
* A participant who experienced an asthma exacerbation that resulted in emergency treatment, hospitalization due to asthma, or treatment with systemic steroids at any time from 1 month prior to Visit 1.
* A participant who had experienced an upper or lower respiratory tract infection within the 4 weeks prior to Visit 1.
* Evidence of lung disease(s) other than asthma.
* Previous smoker (smoking history >10 pack-years) or current smoker (within 6 months prior to Visit 1).
* Comorbid disease that might interfere with the evaluation of investigational medicinal product or conduct of study procedures (e.g., bronchoscopy).
* Anti-immunoglobulin E (IgE) therapy (omalizumab) or any other biologic therapy within 6 months of Visit 1.
* Exposure to another investigative study medication within a time period prior to Visit 1 that is less than 5 half-lives of the study medication.
* Treatment with systemic (oral or injectable) corticosteroids within 28 days of Visit 1.

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2016-01-27 (Actual); Primary Completion 2018-01-03 (Actual); Study Completion 2018-01-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (16):
- United States (6):
  - Investigational Site Number 840402, Tucson, Arizona
  - Investigational Site Number 840403, Denver, Colorado
  - Investigational Site Number 840401, Boston, Massachusetts
  - Investigational Site Number 840002, St Louis, Missouri
  - Investigational Site Number 840404, Winston-Salem, North Carolina
  - Investigational Site Number 840028, Pittsburgh, Pennsylvania
- Canada (2):
  - Investigational Site Number 124012, Montreal
  - Investigational Site Number 124018, Sainte-Foy
- Denmark (2):
  - Investigational Site Number 208002, Hvidovre
  - Investigational Site Number 208001, København NV
- Germany (3):
  - Investigational Site Number 276013, Frankfurt am Main
  - Investigational Site Number 276011, Großhansdorf
  - Investigational Site Number 276012, Hanover
- Investigational Site Number 752001, Lund, Sweden
- United Kingdom (2):
  - Investigational Site Number 826010, London
  - Investigational Site Number 826009, Oxford

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 16 sites in 6 countries. A total of 133 participants were screened between January 2016 and January 2018. Of which, 42 participants were randomized. 91 participants were screen failures mainly due to exclusion criteria met and inclusion criteria not met.
Pre-assignment Details: Participants were randomized in 1:1 ratio to receive dupilumab 300 mg every 2 weeks (q2w) and placebo q2w by using Interactive Voice/Web Response System (IVRS). Randomization was stratified by inhaled corticosteroids (ICS) dose (medium and high) and region (North America and Europe).
Groups:
- Placebo: Placebo (for dupilumab), 2 subcutaneous injections on Day 1 (Week 1) as a loading dose followed by a single injection q2w from Week 2 to Week 14 added to stable inhaled corticosteroid/ long-acting beta-agonist (ICS/LABA) therapy. Salbutamol/albuterol or Levosalbutamol/levalbuterol was given as reliever medication.
- Dupilumab: Dupilumab, 2 subcutaneous injections on Day 1 as a loading dose for a total of 600 mg, followed by a single 300 mg injection q2w from Week 2 to Week 14 added to stable ICS/LABA therapy. Salbutamol/albuterol or Levosalbutamol/levalbuterol was given as reliever medication.
Period: Overall Study
Arm/Group | Placebo | Dupilumab
Started | 22 | 20
Completed | 22 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline population included all randomized participants.
Groups:
- Placebo: Placebo (for dupilumab), 2 subcutaneous injections on Day 1 (Week 1) as a loading dose followed by a single injection q2w from Week 2 to Week 14 added to stable ICS/LABA therapy. Salbutamol/albuterol or Levosalbutamol/levalbuterol was given as reliever medication.
- Total: Total of all reporting groups
Arm/Group | Placebo | Dupilumab | Total
Number analyzed (Participants) | 22 | 20 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.0 (10.3) | 45.5 (10.6) | 43.1 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 13 | 21
  Male | 14 | 7 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 21 | 19 | 40
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 19 | 16 | 35
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Baseline Eosinophils Count in Bronchial Tissue [Median (Inter-Quartile Range); unit: cells/mm^2] — Inflammatory cells i.e. eosinophils were counted in the bronchial submucosa of biopsy thin sections using quantitative immunohistochemistry and reported as the number of cells per square millimeter. Population: Here, number analyzed = participants with available data at baseline.
  cells/mm^2
    number analyzed (Participants) | 21 | 19 | 40
    (all) | 12.97 [9.91 to 21.24] | 34.96 [10.07 to 263.75] | 20.73 [9.99 to 68.87]
Baseline Mucin-Stained Area in The Bronchial Tissue Specimen [Mean (Standard Deviation); unit: cells/mm^2] — Mucin was identified by staining with Alcian-blue periodic acid-Schiff and/or immunostaining for MUC5AC and then the mucin-positive area was measured and expressed per square millimeter. Population: Here, number analyzed = participants with available data at baseline.
  cells/mm^2
    number analyzed (Participants) | 22 | 19 | 41
    (all) | 561.12 (289.00) | 520.57 (511.69) | 542.33 (402.61)
Baseline Mast Cells Count (Chymase Positive) in Bronchial Tissue [Mean (Standard Deviation); unit: cells/mm^2] — Inflammatory cells i.e. mast cells were counted in the bronchial submucosa of biopsy thin sections using quantitative immunohistochemistry and reported as the number of cells per square millimeter.
  cells/mm^2 | 74.36 (58.63) | 79.17 (68.07) | 76.59 (62.42)
Baseline Mast Cells Count (Tryptase Positive) in Bronchial Tissue [Mean (Standard Deviation); unit: cells/mm^2] — Inflammatory cells i.e. mast cells were counted in the bronchial submucosa of biopsy thin sections using quantitative immunohistochemistry and reported as the number of cells per square millimeter. Population: Here, number analyzed = participants with available data at baseline.
  cells/mm^2
    number analyzed (Participants) | 22 | 19 | 41
    (all) | 80.10 (64.92) | 105.53 (104.68) | 91.88 (85.49)
Baseline Total T-Lymphocytes Count in Bronchial Tissue [Median (Inter-Quartile Range); unit: cells/mm^2] — T-Lymphocytes i.e. CD3 positive cells were counted in the bronchial submucosa of biopsy thin sections using quantitative immunohistochemistry and reported as the number of cells per square millimeter. Population: Here, number analyzed = participants with available data at baseline.
  cells/mm^2
    number analyzed (Participants) | 22 | 19 | 41
    (all) | 301.09 [121.01 to 500.43] | 153.33 [83.81 to 192.40] | 181.50 [105.08 to 392.13]
Baseline T-Helper Lymphocytes Count in Bronchial Tissue [Median (Inter-Quartile Range); unit: cells/mm^2] — T-helper i.e. CD4 positive lymphocytes were counted in the bronchial submucosa of biopsy thin sections using quantitative immunohistochemistry and reported as the number of cells per square millimeter. Population: Here, number analyzed = participants with available data at baseline.
  cells/mm^2
    number analyzed (Participants) | 22 | 19 | 41
    (all) | 237.10 [190.17 to 511.48] | 200.85 [102.49 to 398.08] | 215.05 [147.29 to 467.90]
Baseline Fractional exhaled nitric oxide (FeNO) [Mean (Standard Deviation); unit: parts per billion (ppb)] — FeNO is a surrogate marker for airway inflammation. FeNO was analyzed using a NIOX instrument or similar analyzer using a flow rate of 50 mL/s, and reported in ppb.
  parts per billion (ppb) | 41.2 (31.5) | 36.4 (22.8) | 38.9 (27.5)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Eosinophils Cells Count in the Bronchial Submucosa at Week 12
Description: Inflammatory cells i.e. eosinophils were counted in the bronchial submucosa of biopsy thin sections using quantitative immunohistochemistry and reported as the number of cells per square millimeter.
Time Frame: Baseline, Week 12
Population: Analysis was performed on pharmacodynamic (PD) population which consisted of all randomized participants who underwent baseline and Week12/end of treatment (EOT) bronchoscopies and have adequate biopsies for analysis at both baseline and EOT. Here, overall number of participants analyzed = participants with available data for this outcome measure.
Measure: Median (Inter-Quartile Range); unit: cells/mm^2
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 20 | 17
cells/mm^2 | 5.80 [-9.18 to 33.41] | -6.04 [-174.71 to 19.41]
Statistical Analysis 1: Comparison: Placebo vs Dupilumab; Analysis was performed using a rank ANCOVA model stratified by ICS dose level and region; Test type: Superiority; p = 0.8400, Rank ANCOVA — Threshold for significance at 0.05 level; Rank ANCOVA model stratified by ICS dose level and region

2. Primary Outcome: Change From Baseline in Mucin-Stained Area in the Bronchial Submucosa at Week 12
Description: Mucin was identified by staining with Alcian-blue periodic acid-Schiff and/or immunostaining for MUC5AC and then the mucin-positive area was measured and expressed per square millimeter.
Time Frame: Baseline, Week 12
Population: Analysis was performed on PD population. Here, overall number of participants analyzed = participants with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: cells/mm^2
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 20 | 16
cells/mm^2 | 64.09 (391.96) | -142.74 (477.89)
Statistical Analysis 1: Comparison: Placebo vs Dupilumab; Analysis was performed using a linear fixed-effect model with treatment, region and ICS dose level as fixed effects, and the baseline value as continuous covariate; Test type: Superiority; p = 0.0336, Linear fixed-effect model — Threshold for significance at 0.05 level; LS Mean Difference = -235.02, 90% CI 2-sided [-414.19 to -55.84]

3. Primary Outcome: Change From Baseline in Mast Cells Count (Chymase Positive) in the Bronchial Submucosa at Week 12
Description: Inflammatory cells i.e. mast cells were counted in the bronchial submucosa of biopsy thin sections using quantitative immunohistochemistry and reported as the number of cells per square millimeter.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: cells/mm^2
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 20 | 17
cells/mm^2 | -14.80 (76.52) | 1.76 (62.41)
Statistical Analysis 1: Comparison: Placebo vs Dupilumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.4795, Linear fixed-effect model — Threshold for significance at 0.05 level; LS mean difference = 13.89, 90% CI 2-sided [-19.00 to 46.78]

4. Primary Outcome: Change From Baseline in Mast Cells Count (Tryptase Positive) in the Bronchial Submucosa at Week 12
Description: as for outcome 3
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: cells/mm^2
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 21 | 17
cells/mm^2 | 2.37 (90.20) | -20.89 (59.09)
Statistical Analysis 1: Comparison: Placebo vs Dupilumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.4494, Linear fixed-effect model — Threshold for significance at 0.05 level; LS mean difference = -18.98, 90% CI 2-sided [-60.92 to 22.97]

5. Primary Outcome: Change From Baseline in T-Lymphocytes Count in the Bronchial Submucosa at Week 12
Description: T-Lymphocytes i.e. CD3 positive cells were counted in the bronchial submucosa of biopsy thin sections using quantitative immunohistochemistry and reported as the number of cells per square millimeter.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: cells/mm^2
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 20 | 16
cells/mm^2 | -36.70 [-200.25 to 267.51] | 34.21 [-95.08 to 232.99]
Statistical Analysis 1: Comparison: Placebo vs Dupilumab; Analysis was performed using a rank ANCOVA model stratified by ICS dose level and region; Test type: Superiority; p = 0.6865, Rank ANCOVA — Threshold for significance at 0.05 level; Rank ANCOVA model stratified by ICS dose level and region

6. Primary Outcome: Change From Baseline in T-Helper Lymphocytes Count in the Bronchial Submucosa at Week 12
Description: T-helper i.e. CD4 positive lymphocytes were counted in the bronchial submucosa of biopsy thin sections using quantitative immunohistochemistry and reported as the number of cells per square millimeter.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: cells/mm^2
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 20 | 16
cells/mm^2 | 7.26 [-179.43 to 224.96] | 62.34 [-100.62 to 159.09]
Statistical Analysis 1: Comparison: Placebo vs Dupilumab; Analysis was performed using a rank ANCOVA model stratified by ICS dose level and region; Test type: Superiority; p = 0.7588, Rank ANCOVA — Threshold for significance at 0.05 level; Rank ANCOVA model stratified by ICS dose level and region

7. Secondary Outcome: Change From Baseline in Fractional Exhaled Nitric Oxide (FeNO) at Week 12
Description: FeNO is a surrogate marker for airway inflammation. FeNO was analyzed using a NIOX instrument or similar analyzer using a flow rate of 50 mL/second, and reported in ppb.
Time Frame: Baseline, Week 12
Population: Analysis was performed on secondary PD population which consisted of all randomized and treated participants. Here, overall number of participants analyzed = participants with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: ppb
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 21 | 18
ppb | 3.9 (22.8) | -15.1 (18.3)
Statistical Analysis 1: Comparison: Placebo vs Dupilumab; Analysis was performed using a Mixed-effect Model with Repeated Measures (MRMM) with treatment, treatment-by-visit interaction, region, and ICS dose level as fixed effects, and baseline biomarker-by-visit interaction as fixed covariate, and assuming an unstructured covariance structure separately by treatment group; Test type: Superiority; p = 0.0012, MMRM — Threshold for significance at 0.05 level; LS Mean Difference = -22.4, 90% CI 2-sided [-32.9 to -11.9]

8. Secondary Outcome: Average Change in Fractional Exhaled Nitric Oxide (FeNO) From Baseline to Week 6 Through Week 12
Description: FeNO is a surrogate marker for airway inflammation. FeNO was analyzed using a NIOX instrument or similar analyzer using a flow rate of 50 mL/s, and reported in ppb.
  The average change in FeNO from baseline to Week 6 through Week 12 was calculated as follows: For each participant the change in FeNO from Baseline to Week 6, Week 8, Week 10 and Week 12 was calculated (value at Week X - value at baseline). Subsequently the weekly mean of these 4 "change from baseline" values was determined (Weeks 6, 8, 10 and 12). Using these weekly mean values the overall arithmetic mean and standard deviation of the average change in FeNO from baseline to Week 6 through Week 12 was calculated.
Time Frame: From Baseline to Week 6 through Week 12
Population: Analysis was performed on secondary PD population.
Measure: Mean (Standard Deviation); unit: ppb
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 22 | 20
ppb | 3.5 (18.0) | -16.0 (21.0)
Statistical Analysis 1: Comparison: Placebo vs Dupilumab; Analysis was performed using a Mixed-effect model with Repeated Measures (MMRM) with treatment, treatment-by-visit interaction, region, and ICS dose level as fixed effects, and baseline biomarker-by-visit interaction as fixed covariate, and assuming an unstructured covariance structure separately by treatment group; Test type: Superiority; p = 0.0005, MMRM — Threshold for significance at 0.05 level; LS Mean Difference = -22.0, 90% CI 2-sided [-31.3 to -12.8]

9. Secondary Outcome: Number of Participants With Antidrug Antibodies (ADA)
Description: Anti-drug antibodies were detected using a validated immunoassay. Incidence of ADA were classified as following: 1) Pre-existing immunoreactivity - an ADA positive response in the assay at baseline with all post treatment ADA results negative or an ADA positive response at baseline with all post treatment ADA responses less than 4-fold over baseline titer levels. 2) Treatment-emergent ADA: an ADA positive response in the assay post first dose, when baseline results were negative or missing. 3) Treatment-boosted ADA: an ADA positive response in the assay post first dose that was greater-than or equal to 4-fold over baseline titer levels, when baseline results were positive.
Time Frame: From Baseline up to 24 weeks
Population: Analysis was performed on ADA population which consisted of all participants with at least one qualified ADA result in the ADA assay following the first dose of the study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 21 | 19
Participants
  With pre-existing immunoreactivity | 1 | 0
  With treatment-emergent ADA | 0 | 1
  With treatment-boosted ADA | 0 | 0

10. Secondary Outcome: Pharmacokinetics (PK) Assessment: Serum Functional Dupilumab Concentration
Description: Serum functional dupilumab concentrations were determined using an enzyme-linked immunosorbent assay (ELISA) method.
Time Frame: Week 0, Week 2, 6, 8, 12, 18, End of study (Week 24)
Population: Analysis was performed on PK population which consisted of all participants with at least one non-missing and eligible post-baseline dupilumab serum concentration data. Data for this outcome measure was not planned to be analyzed for placebo arm. Here, "number analyzed" represents number of subjects with available data for specified time points.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Dupilumab
Number analyzed (Participants) | 20
ng/mL
  Week 0 | 0.00 (0.00)
  Week 2 | 52675.00 (23107.55)
  Week 6 | 59969.00 (27422.27)
  Week 8 | 61097.95 (29775.23)
  Week 12 | 67387.00 (32800.44)
  Week 18: number analyzed (Participants) | 6
  Week 18 | 20728.17 (17718.93)
  Week 24: number analyzed (Participants) | 5
  Week 24 | 1851.20 (2796.78)

11. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: Adverse event (AE) was defined as any untoward medical occurrence in a participant who received investigational medicinal product (IMP) without regard to possibility of causal relationship with this treatment. TEAEs: AEs that developed or worsened or became serious during between the first administration of study medication to the end of the 12 week Post-treatment Period. Serious adverse event (SAE) was defined as any untoward medical occurrence that resulted in any of the following outcomes: death, life-threatening, required initial or prolonged in-patient hospitalization, persistent or significant disability/incapacity, congenital anomaly/birth defect, or considered as medically important event. Any TEAE included both serious and non-serious AEs.
Time Frame: Baseline up to Week 24
Population: Analysis was performed on safety population which consisted of all participants randomized and exposed to study medication, regardless of the amount of treatment administered.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 22 | 20
Participants
  Any TEAE | 17 | 15
  Any treatment emergent SAE | 0 | 1
  Any TEAE leading to death | 0 | 0
  Any TEAE leading to permanent discontinuation | 0 | 0

ADVERSE EVENTS:
Time Frame: All AEs were collected from signature of the informed consent form up to the end of study (i.e. up to the end of Post-treatment period [Week 24]) regardless of seriousness or relationship to investigational medicinal product (IMP).
Description: Reported AEs and deaths are treatment emergent AEs that developed/worsened and deaths that occurred during 'treatment-emergent period' (from first dose of investigational product injection up to the end of Post-treatment period [Week 24]). Analysis was performed on safety population.
Arm/Group | Placebo | Dupilumab
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/22 | 1/20
Other Adverse Events (participants affected / at risk) | 11/22 | 14/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=22) | Dupilumab (N=20)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=22) | Dupilumab (N=20)
Nausea (Gastrointestinal disorders) | 1 (1) | 3 (3)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2)
Injection Site Erythema (General disorders) | 2 (8) | 3 (8)
Injection Site Inflammation (General disorders) | 2 (3) | 1 (3)
Injection Site Pruritus (General disorders) | 1 (1) | 2 (3)
Nasopharyngitis (Infections and infestations) | 4 (6) | 2 (2)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 3 (3)
Accidental Overdose (Injury, poisoning and procedural complications) | 1 (1) | 2 (3)
Road Traffic Accident (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Headache (Nervous system disorders) | 3 (9) | 5 (11)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 2 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.

DOCUMENTS (2):
  • Study Protocol (2016-11-23): https://cdn.clinicaltrials.gov/large-docs/33/NCT02573233/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-09): https://cdn.clinicaltrials.gov/large-docs/33/NCT02573233/SAP_001.pdf